CLINICAL TRIAL: NCT00553059
Title: Randomized, Double-Blind, Placebo-Controlled Trial of Palonosetron/Dexamethasone With or Without Dronabinol for the Prevention of Chemotherapy-Induced Nausea and Vomiting After Moderately Emetogenic Chemotherapy
Brief Title: Palonosetron and Dexamethasone With or Without Dronabinol in Preventing Nausea and Vomiting in Patients Receiving Chemotherapy For Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Solvay Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2006-0841; MDA-2006-0841; CDR0000573510 (Other: NCI); NCI-2009-00637 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-11-02; First posted 2007-11-05 (Estimated); Results first posted 2020-10-09 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Chemotherapy-induced Nausea and Vomiting; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: nausea and vomiting; unspecified adult solid tumor; Palonosetron; Dexamethasone
MeSH Terms: conditions — Vomiting; Nausea | interventions — Dexamethasone; Dronabinol; Palonosetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I: Palonosetron, Dexamethasone + Dronabinol (Experimental): Palonosetron hydrochloride intravenous (IV) and dexamethasone IV 30 minutes before chemotherapy administration on day 1, and oral dronabinol 3 times a day for 5 days beginning 30 minutes before chemotherapy administration on day 1.
  Interventions: Drug: dexamethasone; Drug: dronabinol; Drug: palonosetron hydrochloride
- Arm II: Palonosetron + Dexamethasone (Active Comparator): Palonosetron hydrochloride and dexamethasone as in arm I, and oral placebo 3 times a day for 5 days beginning 30 minutes before chemotherapy on day 1.
  Interventions: Drug: dexamethasone; Drug: palonosetron hydrochloride; Other: placebo

INTERVENTIONS:
Drug: dexamethasone — 10 mg IV 30 minutes prior to administration of chemotherapy
Drug: dronabinol — 5 mg tablet by mouth three times a day beginning 30 minutes before chemotherapy
  Arms: Arm I: Palonosetron, Dexamethasone + Dronabinol
Drug: palonosetron hydrochloride — 0.25 mg IV 30 minutes prior to administration of chemotherapy
Other: placebo — 1 tablet by mouth three times a day beginning 30 minutes before chemotherapy
  Arms: Arm II: Palonosetron + Dexamethasone

SUMMARY:
The goal of this clinical research study is to learn if adding dronabinol in combination with the standard of care (dexamethasone and palonosetron) can better help to control nausea and vomiting in patients receiving chemotherapy. The safety of the drug combinations will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Dronabinol and palonosetron are both designed to help prevent nausea and vomiting in patients who are receiving chemotherapy.

Dexamethasone is a corticosteroid that is similar to a natural hormone made by your body. Dexamethasone is often given to MM patients in combination with other chemotherapy to treat cancer.

Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 groups.

* If you are in Group 1, you will take dronabinol, dexamethasone, and palonosetron.
* If you are in Group 2, you will take a placebo, dexamethasone, and palonosetron. A placebo is a substance that looks like the study drug but has no active ingredients.

You will have an equal chance of being assigned to either group. Neither you nor your doctor can choose the group you will be in. During the study, you and the study staff will not know which group you are in. However, if needed for your safety, the study staff will be able to find out which group you are in.

After the last study participant completes their study therapy, you and the study staff will find out which group you were in.

Study Drug Administration:

On Day 1 (the day that you receive chemotherapy), you will take a dronabinol/placebo pill by mouth every 8 hours (if possible). If you cannot take the pill every 8 hours, you should try to space out the doses evenly. Your first dronabinol/placebo pill on Day 1 will be 30 minutes before chemotherapy.

You will also receive dexamethasone and palonosetron by vein 30 minutes before you receive chemotherapy.

On Days 2-6, you will take dronabinol/placebo 3 times a day. You should take each pill every 8 hours (if possible). If you cannot take them every 8 hours, you should try to space out the doses evenly.

Study Diary:

You will complete a study diary on Days 1-6. In this diary you will answer questions about nausea and vomiting.

Study Visits:

You will have a study visit on Day 8 and again sometime during Days 14-28. At both visits, you will be asked if you have experienced any side effects. You should return your study diary to the clinic at both visits. At the visit during Days 14-28, you will also have a physical exam.

Length of Study:

You will be on study for 30 days. You will be taken off study early if the nausea and vomiting do not improve or intolerable side effects occur.

This is an investigational study. Dronabinol and palonosetron are both FDA approved and commercially available to prevent nausea and vomiting that may occur from chemotherapy. Dexamethasone is FDA approved and commercially available for the prevention of side effects related to chemotherapy. The combination of these drugs to prevent nausea and vomiting is investigational.

Up to 200 patients will take part in this multicenter study. Up to 200 will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically documented solid tumor
2. Receiving moderately emetogenic chemotherapy for the first time: Patients may be chemotherapy naive, or patients may have previously received a mildly emetogenic agent (such as a taxane) if no nausea/vomiting was experienced with that chemotherapy
3. Scheduled to receive cyclophosphamide </= 1500 mg/m^2 IV and/or doxorubicin >/= 40 mg/m^2 IV given as single doses on Day 1. Patients on combination regimens with these agents are eligible
4. Age >/= 18 years
5. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
6. Adequate organ reserve as follows: 1) Hematologic - white blood cell count (WBC) >/= 3000/microL, AGC >/= 1500/microL, platelet >/= 100,000/microL; 2) Renal - Creatinine </= 1.5 times upper limit of normal; 3) Hepatic - Bilirubin and transaminases </= 2.5 times upper limit of normal
7. The effects of the three-drug regimen on the developing human fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; or abstinence) for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
8. Negative qualitative B-human chorionic gonadotropin (HCG) (pregnancy test)
9. Signed informed consent

Exclusion Criteria:

1. Scheduled to receive highly emetogenic chemotherapy (Hesketh Level 5 - such as cisplatin, streptozotocin, dacarbazine, carmustine, hexamethylmelamine, mechlorethamine, procarbazine) during the study period
2. Scheduled to receive moderately emetogenic chemotherapy (Hesketh Level 3-4) after Day 1 of the study period
3. Experienced nausea and/or vomiting with prior administration of chemotherapy
4. Prior moderately or highly emetogenic chemotherapy: Patients may have previously received a mildly emetogenic agent (such as a taxane) if no nausea/vomiting was experienced with that chemotherapy
5. Scheduled to receive cranial, abdominal, or pelvic radiation therapy during the study period
6. Treatment with any investigational agent within 30 days of randomization
7. Scheduled to receive treatment during the study period with other potential or known antiemetic agents. Chronically used benzodiazepines may be continued as a single nightly dose for sleep.
8. Scheduled to receive corticosteroid treatment other than the study drug dose during the study period
9. Uncontrolled primary or metastatic CNS tumor (including those with uncontrolled seizures)
10. Other physical causes for nausea or vomiting (such as bowel obstruction) not related to chemotherapy administration
11. Recent history of unexplained nausea or vomiting or history of frequent nausea or vomiting
12. Active bacterial or fungal infection for which administration of a corticosteroid would be contraindicated
13. Hypersensitivity to any of the study agents
14. Sensitivity to sesame oil
15. Planned simultaneous administration of any other investigational agents
16. Pregnant or nursing women
17. Previous poor tolerance of cannabinoids
18. Habitual cannabinoid use or unwillingness to avoid the use of marijuana during the study period
19. Previous use of dronabinol or nabilone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2008-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven M. Grunberg, MD, Study Chair — University of Vermont; Amal I. Melhem-Bertrandt, MD, Study Chair — M.D. Anderson Cancer Center
Locations (4):
- United States (4):
  - Cancer Research for the Ozarks, Springfield, Missouri
  - CCOP - Greenville, Greenville, South Carolina
  - University of Texas M.D. Anderson, Houston, Texas
  - Vermont Cancer Center at University of Vermont, Burlington, Vermont

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: May 13, 2008 to October 26, 2011. Recruitment done in various medical clinics.
Groups:
- Dronabinol: Dronabinol 1 capsule three times per day for 5 days
- Placebo: Placebo 1 capsule three times per day for 5 days
Period: Overall Study
Arm/Group | Dronabinol | Placebo
Started | 31 | 31
Completed | 30 | 29
Not Completed | 1 | 2
Not completed — Deemed ineligible | 1 | 1
Not completed — Drug supply not available | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dronabinol | Placebo | Total
Number analyzed (Participants) | 31 | 31 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 19 | 37
  >=65 years | 13 | 12 | 25
Age, Continuous [Median (Full Range); unit: years] | 59 [37 to 75] | 57 [29 to 76] | 58 [29 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 30 | 61
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 30 | 30 | 60
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 8 | 14
  White | 25 | 22 | 47
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 31 | 31 | 62
Daily Assessment of Nausea and Vomiting [Count of Participants; unit: Participants] — To determine whether dronabinol can add significantly to the antiemetic protection provided by a standard palonosetron and dexamethasone regimen for patients receiving moderately emetogenic chemotherapy.
  Participants | 30 | 29 | 59

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Total Protection in the Acute, Delayed and Overall Periods
Description: Total protection is defined as no vomiting, no rescue therapy, and no nausea as indicated by responses to the acute (0-24 hour), delayed (24-120 hour), and overall (0-120 hour) periods as indicated by responses to the Daily Assessment of Nausea and Vomiting questionnaire. Data to be recorded in the study diary during the 5-day study period. The assessment measures in detail the occurrence, duration, and severity of post-chemotherapy nausea and emesis using a 10-point Likert-type scale ranging from 0 (none) to 10 (as bad as it could be) if nausea or vomiting is present.
Time Frame: 5 Days (first 5 days of the first cycle of chemotherapy)
Measure: Count of Participants; unit: Participants
Arm/Group | Dronabinol | Placebo
Number analyzed (Participants) | 31 | 31
Participants
  Acute | 22 | 14
  Delayed | 11 | 5
  Overall | 11 | 5

2. Secondary Outcome: Number of Participants With Complete Protection for the Acute, Delayed, and Overall Periods
Description: Complete Protection is no vomiting, no rescue therapy, and no nausea evaluated for the acute (0-24 hour), delayed (24-120 hour), and overall (0-120 hour) periods as indicated by responses to the Daily Assessment of Nausea and Vomiting questionnaire. The assessment measures in detail the occurrence, duration, and severity of post-chemotherapy nausea and emesis using a 10-point Likert-type scale ranging from 0 (none) to 10 (as bad as it could be) if nausea or vomiting is present.
Time Frame: Up to 5 days (first 5 days following first cycle of chemotherapy)
Measure: Count of Participants; unit: Participants
Arm/Group | Dronabinol | Placebo
Number analyzed (Participants) | 30 | 29
Participants
  Acute | 22 | 18
  Delayed | 14 | 10
  Overall | 14 | 9

3. Secondary Outcome: Number of Participants With Complete Response for the Acute, Delayed, and Overall Periods
Description: Complete response is defined as vomiting episodes with rescue medication evaluated for the acute (0-24 hour), delayed (24-120 hour), and overall (0-120 hour) periods as indicated by responses to the Daily Assessment of Nausea and Vomiting questionnaire. The assessment measures in detail the occurrence, duration, and severity of post-chemotherapy nausea and emesis using a 10-point Likert-type scale ranging from 0 (none) to 10 (as bad as it could be) if nausea or vomiting is present.
Time Frame: Up to 5 days (first 5 days following first cycle of chemotherapy)
Measure: Count of Participants; unit: Participants
Arm/Group | Dronabinol | Placebo
Number analyzed (Participants) | 30 | 29
Participants
  Acute | 22 | 19
  Delayed | 14 | 13
  Overall | 15 | 12

4. Secondary Outcome: Number of Participants With Vomiting for the Acute, Delayed and Overall Periods
Description: Number of Participants with Vomiting Acute, Delayed and Overall. Evaluated for the acute (0-24 hour), delayed (24-120 hour), and overall (0-120 hour) periods as indicated by responses to the Daily Assessment of Nausea and Vomiting questionnaire. The assessment measures in detail the occurrence, duration, and severity of post-chemotherapy nausea and emesis using a 10-point Likert-type scale ranging from 0 (none) to 10 (as bad as it could be) if nausea or vomiting is present.
Time Frame: 5 Days (first 5 days of the first cycle of chemotherapy)
Measure: Count of Participants; unit: Participants
Arm/Group | Dronabinol | Placebo
Number analyzed (Participants) | 30 | 19
Participants
  Acute | 6 | 3
  Delayed | 10 | 9
  Overall | 19 | 19

5. Secondary Outcome: Number of Participants With Nausea for the Acute, Delayed and Overall Periods
Description: Number of Participants with Nausea for the Acute, Delayed and Overall Periods. Evaluated for the acute (0-24 hour), delayed (24-120 hour), and overall (0-120 hour) periods as indicated by responses to the Daily Assessment of Nausea and Vomiting questionnaire. The assessment measures in detail the occurrence, duration, and severity of post-chemotherapy nausea and emesis using a 10-point Likert-type scale ranging from 0 (none) to 10 (as bad as it could be) if nausea or vomiting is present.
Time Frame: 5 Days (first 5 days of the first cycle of chemotherapy)
Measure: Count of Participants; unit: Participants
Arm/Group | Dronabinol | Placebo
Number analyzed (Participants) | 30 | 29
Participants
  Acute | 8 | 15
  Delayed | 19 | 23
  Overall | 11 | 5

6. Secondary Outcome: Number of Participants With Nausea and Vomiting for the Acute, Delayed and Overall Periods
Description: Number of Participants With Nausea and Vomiting for the Acute, Delayed and Overall Periods. Evaluated for the acute (0-24 hour), delayed (24-120 hour), and overall (0-120 hour) periods as indicated by responses to the Daily Assessment of Nausea and Vomiting questionnaire. The assessment measures in detail the occurrence, duration, and severity of post-chemotherapy nausea and emesis using a 10-point Likert-type scale ranging from 0 (none) to 10 (as bad as it could be) if nausea or vomiting is present.
Time Frame: 5 Days (first 5 days of the first cycle of chemotherapy)
Measure: Count of Participants; unit: Participants
Arm/Group | Dronabinol | Placebo
Number analyzed (Participants) | 30 | 29
Participants
  Acute | 4 | 2
  Delayed | 7 | 8
  Overall | 15 | 10

7. Secondary Outcome: Number of Participants Received Rescue Medication in the Acute, Delayed and Overall Periods
Description: The assessment measures in detail the occurrence, duration, and severity of post-chemotherapy nausea and emesis using a 10-point Likert-type scale ranging from 0 (none) to 10 (as bad as it could be) if nausea or vomiting is present. The first section asks the patient to record presence and severity of nausea during the last 24 hours. The second section asks the patient to record vomiting episodes during the last 24 hours. The third section asks if the patient took medication for nausea or vomiting during the last 24 hours and asks how useful the treatment for nausea or vomiting was. The fourth section screens for toxicity by asking about side effects and problems experienced during the last 24 hours. Use of rescue antiemetic medication and adverse events also assessed and documented.
Time Frame: 5 Days (first 5 days of the first cycle of chemotherapy)
Measure: Count of Participants; unit: Participants
Arm/Group | Dronabinol | Placebo
Number analyzed (Participants) | 30 | 29
Participants
  Acute | 3 | 5
  Delayed | 11 | 15
  Response | 10 | 12

ADVERSE EVENTS:
Time Frame: 2 years, 8 months
Description: An adverse event (AE) is any condition that appears or worsens after the subject is enrolled in an investigational study. AEs will be graded by numerical score according to the NCI Common Terminology Criteria Adverse Events (CTCAE) version 4.0.
Arm/Group | Dronabinol | Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/29
Serious Adverse Events (participants affected / at risk) | 1/30 | 1/29
Other Adverse Events (participants affected / at risk) | 26/30 | 25/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dronabinol (N=30) | Placebo (N=29)
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Dehydration (Gastrointestinal disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dronabinol (N=30) | Placebo (N=29)
Anemia (Blood and lymphatic system disorders) | 3 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 2 | 0
Other (Blood and lymphatic system disorders) | 7 | 11
Chest Pain (Cardiac disorders) | 1 | 1
Palpitations (Cardiac disorders) | 0 | 1
Blurred Vision (Eye disorders) | 1 | 0
Conjuctivitis (Eye disorders) | 0 | 1
Watering (Eye disorders) | 1 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 14 | 11
Diarrhea (Gastrointestinal disorders) | 13 | 6
Dry Mouth (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 2
Esophagitis (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0
Mucositis - Oral (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 26 | 25
Oral Pain (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 11 | 11
Other (Gastrointestinal disorders) | 16 | 12
Chills (General disorders) | 1 | 3
Edema - Limbs (General disorders) | 0 | 1
Fatigue (General disorders) | 17 | 11
Fever (General disorders) | 1 | 1
Flu-Like Symptoms (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 1 | 0
Pain (General disorders) | 4 | 2
Other (General disorders) | 4 | 1
Allergeric Reaction (Immune system disorders) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 2
Other (Infections and infestations) | 0 | 1
Other (Injury, poisoning and procedural complications) | 2 | 0
Alanine Aminotransferase Increase (Investigations) | 1 | 1
Alkaline Phosphatase Increase (Investigations) | 2 | 0
Asparate Aminotransferase Increase (Investigations) | 1 | 1
INR Increase (Investigations) | 2 | 0
Neutrophil Count Decrease (Investigations) | 3 | 0
Platelet Count Decrease (Investigations) | 4 | 1
WBC Decrease (Investigations) | 5 | 2
Other (Investigations) | 0 | 6
Anorexia (Metabolism and nutrition disorders) | 7 | 8
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Glucose intolerance (Metabolism and nutrition disorders) | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 2
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1
Other (Metabolism and nutrition disorders) | 3 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 7 | 2
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 3
General Muscle Weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 | 1
Other (Musculoskeletal and connective tissue disorders) | 4 | 3
Concentration Impairment (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 14 | 7
Dysgeusia (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 16 | 16
Hypersomnia (Nervous system disorders) | 0 | 2
Lethargy (Nervous system disorders) | 1 | 1
Paresthesia (Nervous system disorders) | 2 | 0
Somnolence (Nervous system disorders) | 5 | 3
Other (Nervous system disorders) | 1 | 4
Agitation (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 2
Euphoria (Psychiatric disorders) | 3 | 4
Insomnia (Psychiatric disorders) | 15 | 4
Other (Psychiatric disorders) | 2 | 2
Urinary Retention (Renal and urinary disorders) | 2 | 0
Reproductive & Breast (General disorders) | 1 | 0
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dry Skin (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Other (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 3
Nail Loss (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 1 | 0
Scalp Pain (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Ulceration (Skin and subcutaneous tissue disorders) | 1 | 0
Other (Skin and subcutaneous tissue disorders) | 5 | 1
Hot Flashes (Vascular disorders) | 1 | 0
Other (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No